CLINICAL TRIAL: NCT00484367
Title: Family and Group Therapies for Adolescent Alcohol Abuse
Brief Title: A Comparison of Adolescent Group Therapy and Transitional Family Therapy for Adolescent Alcohol and Drug Abusers
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: The Morton Center, Inc. (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Morris D. Stanton, PhD, The Morton Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NIAAA-STA12178; R01AA012178 (NIH); NIH Grant R01 AA12178
Record Dates: First submitted 2007-06-07; First posted 2007-06-08 (Estimated); Last update posted 2011-08-26 (Estimated); Status verified 2008-11

CONDITIONS: Alcohol Abuse; Alcohol Dependence; Cannabis Abuse; Cannabis Dependence; Other Substance Abuse
Keywords: Alcohol abuse; Substance abuse; Cannabis abuse; Adolescents; Group therapy; Family therapy
MeSH Terms: conditions — Alcoholism; Marijuana Abuse; Substance-Related Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 AGT (Active Comparator)
  Interventions: Behavioral: Adolescent group therapy
- 2 TFT (Active Comparator)
  Interventions: Behavioral: Transitional family therapy

INTERVENTIONS:
Behavioral: Adolescent group therapy — Adolescent group therapy
  Arms: 1 AGT
Behavioral: Transitional family therapy — Transitional family therapy
  Arms: 2 TFT

SUMMARY:
The purpose of this study is to compare the effectiveness of two psychosocially-based, manual-driven, behavioral modalities. One of these is a standardized version of the established modality of Adolescent Group Therapy (AGT), which includes both psychoeducational and therapeutic components. The other is a state-of-the-art family therapy approach, Transitional Family Therapy (TFT), which integrates management of the current problem with exploration of multigenerational issues. Both approaches have been developed to expressly target adolescent alcohol problems.

DETAILED DESCRIPTION:
Despite well-founded societal concerns over the use of illicit drugs by youth, alcohol use has persisted for decades as the number one adolescent substance abuse problem in the U.S. Further, research has shown that the earlier the onset of alcohol use, the more likely is a person to develop alcohol dependence later, during adulthood. Consequently, the need is clear for interventions which will arrest this process at the earliest point possible. Hence, interventions that mobilize a youth's social systems to help that young person deal with the problem, i.e., the family and peer systems, would make sense from a number of standpoints. Two primary modalities developed to deal with such issues are those examined here: family therapy and group therapy.

The participants were males and females, ages 13-17 at intake, with a DSM-IV diagnosis of either alcohol abuse or alcohol dependence. Following random assignment to condition, basic treatment in both conditions was based on a 12-session model and took approximately 3-4 months, followed by 1-2 aftercare sessions over an additional 1-2 months. The treatment was provided by therapists who were already working within the community (as opposed, for instance, to graduate students). Follow-up assessments were obtained at 3 months post-treatment, 1 year post-treatment, and 2 years post-treatment, thus allowing determination of the extent to which treatment effects "held up" to a degree not attained by most of the previous outcome studies within this domain.

Comparisons: AGT and TFT are being compared on the extent to which their participants used alcohol, as well as other substances, during the three post-treatment periods. Other comparisons include school performance (grade point average), family relations/functioning, and involvement with the legal system.

ELIGIBILITY:
Inclusion Criteria:

* Male and female outpatients 13-17 years of age at intake.
* Participants had a current DSM-IV diagnosis of either alcohol abuse or alcohol dependence.
* Participants signed a witnessed informed consent.
* Parent or custodian of each (adolescent) participant signed a witnessed informed consent.

Exclusion Criteria:

* Participants who met current DSM-IV criteria for bipolar disorder, psychotic disorder, or eating disorder.
* Enrollment in a residential substance abuse treatment program within 2 months prior to intake.

Ages: 13 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 120 (Actual)
Dates: Start 1999-07; Primary Completion 2012-08 (Estimated); Study Completion 2012-08 (Estimated)

PRIMARY OUTCOMES:
Alcohol use Cannabis use Other substance use | Baseline, 3 months post-treatment, 1 year post-treatment, and 2 years post-treatment

CONTACTS AND LOCATIONS:
Overall Officials: Morris D. Stanton, PhD, Principal Investigator — The Morton Center
Locations (1):
- The Morton Center, Louisville, Kentucky, United States